CLINICAL TRIAL: NCT00003335
Title: A Pilot Study of Unrelated Umbilical Cord Blood Transplantation in Patients With High Risk Hematologic Malignancies
Brief Title: Umbilical Cord Blood Transplantation in Treating Patients With High-Risk Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU4Y97; P30CA043703 (NIH); NCI-G98-1429; CWRU4Y97 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Anemia, Refractory, with Excess of Blasts; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Antilymphocyte Serum; Busulfan; Cyclosporine; Melphalan; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin — antithymocyte globulin IV for three days on days -3 to -1
Drug: busulfan — If TBI is not tolerated, busulfan is substituted and administered orally every 6 hours for 4 days on days -8 to -5.
Drug: cyclosporine — Cyclosporine begin on day -2 and continue for 6 months.
Drug: melphalan — melphalan IV for three days on days -4 to -2
Drug: methylprednisolone — Methylprednisolone IV for three days on days -3 to -1. Methylprednisolone begin on day -2 and continue for 6 months.
Procedure: umbilical cord blood transplantation — On day 0, patients receive umbilical cord blood infusion.
Radiation: radiation therapy — 9 fractions of total body irradiation (TBI) on days -9 to -5

SUMMARY:
RATIONALE: Umbilical cord blood transplantation may allow doctors to give higher doses of chemotherapy or radiation therapy and kill more cancer cells.

PURPOSE: This phase II trial is studying allogeneic umbilical cord blood transplantation to see how well it works when given with chemotherapy or radiation therapy in treating patients with high-risk hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rates of hematologic and immune reconstitution in patients with high risk hematologic malignancies who are undergoing high dose chemoradiotherapy followed by unrelated umbilical cord blood (UCB) transplantation.
* Determine the incidence of graft-versus-host-disease in this setting.
* Describe the incidence of recurrent disease in these patients post UCB transplant.
* Describe the incidence of serious infections and secondary lymphoproliferative diseases following transplantation with UCB in these patients.
* Determine specifically whether larger recipients can be durably engrafted with unrelated UCB, and determine whether nucleated cell or progenitor cell content of the graft is predictive of hematological engraftment.

OUTLINE: Patients may undergo a back-up peripheral blood stem cell collection prior to treatment.

Patients receive 9 fractions of total body irradiation (TBI) on days -9 to -5 followed by melphalan IV for three days on days -4 to -2 and antithymocyte globulin IV or methylprednisolone IV for three days on days -3 to -1. On day 0, patients receive umbilical cord blood infusion. If TBI is not tolerated, busulfan is substituted and administered orally every 6 hours for 4 days on days -8 to -5. Cyclosporine and methylprednisolone begin on day -2 and continue for 6 months.

Patients are followed at least monthly for 1 year, then every 6 months for the second year, and then annually thereafter.

PROJECTED ACCRUAL: There will be a maximum of 48 patients accrued into this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high risk malignancy including:

  * Acute nonlymphocytic leukemia (ANLL) after induction failure, or in first complete remission with high risk features including stem cell or biphenotypic classification (acute myeloid leukemia (AML) M0), erythroleukemia (AML M6), acute megakaryocytic leukemia (AML M7), cytogenic markers indicative of poor prognosis, or failure to achieve complete remission after standard induction therapy
  * Acute lymphocytic leukemia (ALL) or ANLL in second or subsequent remission
  * Chronic myeloid leukemia (CML) in chronic phase

    * CML with accelerated phase or blast crisis are eligible after reinduction chemotherapy converts disease to chronic phase
  * High risk ALL in first complete remission
  * Myelodysplastic syndrome with evidence of evolution to acute myeloid leukemia

    * Refractory anemia with excess blasts
    * Refractory anemia with excess blasts in transformation
  * Non-Hodgkin's lymphoma (NHL), ANLL, or ALL with recurrent disease after autologous stem cell transplantation
* Must also meet all the following conditions:

  * No HLA-ABC/DR identical related bone marrow or UCB donor
  * No 5/6 antigen matched related bone marrow or UCB donor
  * Condition precludes waiting to search and find a donor in the National Marrow Donor Registry
* Must have an available serologic matched umbilical cord blood unit in the New York Blood Center's Placental Blood Project
* No active CNS disease

PATIENT CHARACTERISTICS:

Age:

* Under 55 at time of umbilical cord blood transplantation

Performance status:

* Zubrod 0-1
* Karnofsky 80-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* For patients with ALL or ANLL in remission, CML in chronic phase, or NHL without marrow involvement who elect to undergo autologous peripheral blood stem cell collection and storage:

  * WBC at least 3,000/mm^3
  * Absolute neutrophil count at least 1,000/mm^3
  * Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT/AST no greater than 4 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* Normal cardiac function by echocardiogram or radionuclide scan (shortening fraction or ejection fraction at least 80% of normal value for age)

Pulmonary:

* FVC and FEV_1 at least 60% of predicted for age
* For adults:

  * DLCO at least 60% of predicted

Other:

* HIV negative
* No active infections at time of autologous stem cell harvest or pretransplant cytoreduction
* Not pregnant or nursing
* Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior autologous stem cell transplantation allowed

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 1998-01; Primary Completion 2007-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
rates of durable engraftment in patients | day 42
  The primary study end point will be hematologic engraftment. Engraftment is defined as achieving ANC larger than or equal to 500 ul/mm3 of donor origin for three consecutive measurements on different days by day +42.

SECONDARY OUTCOMES:
Event-free survival by clinical and pathological disease assessment | at disease progression or death
incidence of recurrent disease in patients post UCB transplant | post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Brenda W. Cooper, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Lesniewski ML, Haviernik P, Weitzel RP, Kadereit S, Kozik MM, Fanning LR, Yang YC, Hegerfeldt Y, Finney MR, Ratajczak MZ, Greco N, Paul P, Maciejewski J, Laughlin MJ. Regulation of IL-2 expression by transcription factor BACH2 in umbilical cord blood CD4+ T cells. Leukemia. 2008 Dec;22(12):2201-7. doi: 10.1038/leu.2008.234. Epub 2008 Sep 4. PMID 18769450
- [Result] van Heeckeren WJ, Fanning LR, Meyerson HJ, Fu P, Lazarus HM, Cooper BW, Tse WW, Kindwall-Keller TL, Jaroscak J, Finney MR, Fox RM, Solchaga L, Forster M, Creger RJ, Laughlin MJ. Influence of human leucocyte antigen disparity and graft lymphocytes on allogeneic engraftment and survival after umbilical cord blood transplant in adults. Br J Haematol. 2007 Nov;139(3):464-74. doi: 10.1111/j.1365-2141.2007.06824.x. PMID 17910637
- [Derived] Kindwall-Keller TL, Hegerfeldt Y, Meyerson HJ, Margevicius S, Fu P, van Heeckeren W, Lazarus HM, Cooper BW, Gerson SL, Barr P, Tse WW, Curtis C, Fanning LR, Creger RJ, Carlson-Barko JM, Laughlin MJ. Prospective study of one- vs two-unit umbilical cord blood transplantation following reduced intensity conditioning in adults with hematological malignancies. Bone Marrow Transplant. 2012 Jul;47(7):924-33. doi: 10.1038/bmt.2011.195. Epub 2011 Oct 17. PMID 22002488
- [Derived] Weitzel RP, Lesniewski ML, Haviernik P, Kadereit S, Leahy P, Greco NJ, Laughlin MJ. microRNA 184 regulates expression of NFAT1 in umbilical cord blood CD4+ T cells. Blood. 2009 Jun 25;113(26):6648-57. doi: 10.1182/blood-2008-09-181156. Epub 2009 Mar 13. PMID 19286996